CLINICAL TRIAL: NCT04297137
Title: Comparing the Bioavailability of the Sustainable, Non-animal Derived Protein Sources Mycoprotein, Spirulina, Chlorella, Pea and Lupin to Milk Protein in Healthy Older Adults
Brief Title: The Bioavailability of Multiple Novel, Sustainable, Non-animal Derived Protein Sources
Acronym: NOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 191023/A/09
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Healthy Aging
Keywords: Protein digestion; Amino acid absorption; Bioavailability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Mycoprotein (Experimental): Ingestion of 30 g mycoprotein drink
  Interventions: Dietary Supplement: Protein ingestion
- Spirulina (Experimental): Ingestion of 30 g spirulina protein drink
  Interventions: Dietary Supplement: Protein ingestion
- Chlorella (Experimental): Ingestion of 30 g chlorella protein drink
  Interventions: Dietary Supplement: Protein ingestion
- Pea (Experimental): Ingestion of 30 g pea protein drink
  Interventions: Dietary Supplement: Protein ingestion
- Lupin (Experimental): Ingestion of 30 g lupin protein drink
  Interventions: Dietary Supplement: Protein ingestion
- Milk (Active Comparator): Ingestion of 30 g milk protein
  Interventions: Dietary Supplement: Protein ingestion

INTERVENTIONS:
Dietary Supplement: Protein ingestion — Ingestion of various sustainable non-animal derived protein sources compared to animal-based milk protein.

SUMMARY:
The progressive age-related loss of muscle mass is termed sarcopenia. Consequences of sarcopenia are, but not limited to, decreased muscle strength, frailty, and an increased risk for the development of chronic metabolic diseases. Impaired postprandial protein digestion and amino acid absorption with advancing age has been suggested to be a key mechanism underlying sarcopenia. To overcome age-related skeletal muscle atrophy, sufficient dietary protein intake is required. However, the production of animal-based protein sources, such as milk, is associated with a number of economic, environmental, and ethical issues. Accordingly, there is a need to develop sustainable dietary protein sources to support our nutrition. Mycoprotein, spirulina, chlorella, pea, and lupin are novel, sustainable, non-animal derived protein sources that may represent potential alternative protein sources. However, the efficacy of these sources to stimulate muscle mass growth in both young and older adults is unknown.

Therefore, the present study will investigate the postprandial bioavailability of mycoprotein, spirulina, chlorella, pea, and lupin protein when compared to the animal-derived milk protein. Moreover, postprandial protein handling of these novel protein sources across different ages will be assessed. Briefly, 12 healthy young, and older adults will visit the University for 6 separate test days, with each day lasting 6 hours. Participants will consume the one of the 6 protein drinks on each test day. Repeated blood sampling will be used to assess protein digestion and subsequent systemic amino acid appearance.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-35 or 55 - 80 years old.
* Body mass index between 18.5 - 30.

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes).
* Any diagnosed cardiovascular disease or hypertension.
* Elevated blood pressure (>150/90 mmHg) at the time of screening.
* Known pre-existing liver disease/condition.
* Any medication known to affect protein and/or amino acid metabolism.
* Allergy to mycoprotein/Quorn/edible fungi, edible algae, lupin/legumes, or milk.
* Smoking.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Plasma amino acid concentrations | 5 hours
  Peak and total plasma amino acid concentrations following protein ingestion

SECONDARY OUTCOMES:
Blood glucose | 5 hours
  The levels of glucose in the blood following protein ingestion
Serum insulin | 5 hours
  The levels of insulin in blood serum following protein ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Wall, PhD, Principal Investigator — Professor of Nutritional Physiology
Locations (1):
- University of Exeter, Exeter, United Kingdom